CLINICAL TRIAL: NCT02052466
Title: Prediction of Development of Scapular Notching Based on Glenosphere Positioning, Scapular Morphology, and Simulated Impingement-free Motion Using Three-dimensional Computed Tomography Analysis
Brief Title: Prediction of Development of Scapular Notching Following Reverse Total Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Eric Ricchetti (Other)
Responsible Party: Sponsor-Investigator, Eric Ricchetti, Staff, Orthopaedic Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 12-1244
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Rotator Cuff Tear Arthropathy; Reverse Total Shoulder Arthroplasty; Scapular Notching
Keywords: Shoulder Joint; Computed tomography
MeSH Terms: conditions — Osteoarthritis; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reverse TSA patients: Patients having undergone reverse TSA at the Cleveland Clinic with a high quality preoperative CT of the operative shoulder and who are at least 24 months post surgery.

SUMMARY:
The hypothesis is that computer simulated bony impingement of the bone surrounding the spherical glenoid implant (the glenosphere) along the scapular neck on three-dimensional (3-D) computed tomography (CT) imaging analysis is predictive of the location of clinical scapular notching that develops following reverse total shoulder arthroplasty (TSA).

DETAILED DESCRIPTION:
The Specific Aims are:

* Determine the relationship between lateral glenoid offset and the development of scapular notching following reverse TSA
* Determine the ability of 3-D preoperative planning tools to define areas of scapular bony impingement on kinematic simulated shoulder range of motion that predict the development of scapular notching
* Compare the precision and accuracy of plain radiographs (2-D) versus CT (3-D) for measurement of scapular notching and postoperative implant position following reverse TSA (2-D versus 3-D)
* Determine the implant and anatomic factors that best correlate with clinical outcome following reverse TSA by retrospective analysis

ELIGIBILITY:
Inclusion Criteria:

* All patients having undergone reverse TSA at the Cleveland Clinic with a high quality preoperative CT of the operative shoulder and a minimum of two years out from surgery

Exclusion Criteria:

* All patients having undergone reverse TSA at the Cleveland Clinic with no preoperative CT or a low quality preoperative CT of the operative shoulder and/or less than two years from surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had a reverse Total Shoulder Arthroplasty at the Cleveland Clinic from 2004 to 2011 and who had a high quality preoperative CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric T Ricchetti, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iannotti JP, Ricchetti ET, Rodriguez EJ, Bryan JA. Development and validation of a new method of 3-dimensional assessment of glenoid and humeral component position after total shoulder arthroplasty. J Shoulder Elbow Surg. 2013 Oct;22(10):1413-22. doi: 10.1016/j.jse.2013.01.005. Epub 2013 Mar 6. PMID 23473609

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reverse TSA Patients
Started | 32
Completed | 30
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Acromial fracture | 1

BASELINE CHARACTERISTICS:
Groups:
- Reverse TSA Patients: Patients having undergone reverse Total Shoulder Arthroplasty (TSA) at the Cleveland Clinic with a high quality preoperative CT of the operative shoulder and who are at least 24 months post surgery.
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.08 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Actual Versus Predicted Scapular Notching
Description: At minimum 2 year follow-up, compare presence of scapular notching as assessed by 2D x-ray and 3D CT imaging with predicted scapular notching as assessed by 3D computer modeling using video motion analysis of subject range of motion.
Time Frame: At least 24 months after reverse TSA
Population: Patients who had video motion analysis of their range of motion at minimum 2 year follow-up
Measure: Number; unit: percentage of accurate predictions
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 29
percentage of accurate predictions | 96.6

2. Secondary Outcome: Patient Reported Pain, Satisfaction and Function (Penn Shoulder Score)
Description: The Penn Shoulder Score is a shoulder-specific patient reported outcome measure. Best possible score is 100; worst possible score is 0. There are 3 sub-scores: pain (3 questions, 30 possible points), satisfaction (1 question, 10 possible points), and function (20 questions, 60 possible points). Total score is the sum of the 3 sub-scores. For all sub-scores, higher is better.
  The pain questions are based on a 10-point numeric rating scale. Points are added for the pain sub-score.
  The satisfaction question asks the patient to rate their satisfaction with their shoulder. It is based on a 10-point numeric rating scale, with 0 as "not satisfied" and 10 as "very satisfied".
  The function sub-score has 20 questions concerning activities of daily living. The response options are: 0 (can't do at all), 1 (can do with much difficulty), 2 (can do with some difficulty) and 3 (can do with no difficulty). If all activities can be done without difficulty, a score of 60 is achieved.
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Scores on the Penn Shoulder Score scale
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Scores on the Penn Shoulder Score scale | 78.4 (17.2)

3. Secondary Outcome: Shoulder Strength - Flexion
Description: Muscle strength test will be performed three times with each motion and recorded, using the Lafayette Manual Muscle Test System (Model # 01163). Units of output are pounds.
Time Frame: At least 24 months after TSA
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
pounds | 10.2 (3.8)

4. Secondary Outcome: Shoulder Strength - Abduction
Description: as for outcome 3
Time Frame: At least 24 months after TSA
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
pounds | 11.3 (3.8)

5. Secondary Outcome: Shoulder Strength - Internal Rotation
Description: as for outcome 3
Time Frame: At least 24 months after TSA
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
pounds | 9.7 (4.0)

6. Secondary Outcome: Shoulder Strength - External Rotation
Description: as for outcome 3
Time Frame: At least 24 months after TSA
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
pounds | 7.5 (3.2)

7. Secondary Outcome: Active Shoulder Range of Motion - Flexion
Description: Flexion
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 134.5 (27.3)

8. Secondary Outcome: Active Shoulder Range of Motion - Abduction
Description: Abduction
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 120.5 (26.1)

9. Secondary Outcome: Active Shoulder Range of Motion - External Rotation
Description: External rotation
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 26.8 (19)

10. Secondary Outcome: Passive Shoulder Range of Motion - Flexion
Description: Flexion
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 141.7 (24.0)

11. Secondary Outcome: Passive Shoulder Range of Motion - Abduction
Description: Abduction
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 128.0 (25.1)

12. Secondary Outcome: Passive Shoulder Range of Motion - External Rotation
Description: External rotation
Time Frame: At least 24 months after reverse TSA
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Reverse TSA Patients
Number analyzed (Participants) | 30
Degrees | 43 (16.2)

ADVERSE EVENTS:
Time Frame: Minimum 2 years after surgery
Arm/Group | Reverse TSA Patients
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reverse TSA Patients (N=30)
Hip fracture due to fall (Musculoskeletal and connective tissue disorders) | 2 (2) — Treated surgically with hip hemiarthroplasty
Fracture of acromion (Musculoskeletal and connective tissue disorders) | 1 (1) — Minimally displaced fracture of acromion due to motor vehicle accident. Treated surgically with Open Reduction, Internal Fixation.
A-fib with rapid ventricular response (Cardiac disorders) | 1 (1)
Transient ischemic attack (Cardiac disorders) | 1 (1)
Bladder tumor (Renal and urinary disorders) | 1 (1) — Transurethral bladder resection
Pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) — Lower extremity cellulitis
External artery, common femoral, and profunda endarterectomy (Vascular disorders) | 1 (1) — Peripheral vascular disease with lymphoma and claudication
Thiamine deficiency (Metabolism and nutrition disorders) | 1 (1) — Altered mental state

LIMITATIONS AND CAVEATS:
Relatively small sample size. Range of motion was measured at minimum 2 year follow-up, not pre-operatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No